CLINICAL TRIAL: NCT06955351
Title: Survey of Willingness of Police Force in New Taipei City to Participate in Prehospital Resuscitation
Brief Title: REsuscitation Survey of Police Officers in New Taipei City for Duty
Acronym: RESPOND
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: New Taipei City Police Department (Unknown); New Taipei City Fire Department (Unknown)
Responsible Party: Sponsor
Other Study IDs: 112212-E; FEMH-2023-C-046 (Other: Far Eastern Memorinal Hospital)
Record Dates: First submitted 2025-04-15; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Bystander; Chest Compression; Out of Hospital Cardiac Arrest; AED; Police; Willingness to Participate
Keywords: Out-of-Hospital Cardiac Arrest (OHCA); police; Willingness; AED; CPR
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frontline Police Officers in New Taipei City: Frontline police officers in New Taipei City are responsible for various field duties, including patrolling, responding to emergency calls, conducting security checks, traffic control, and maintaining public order. These officers often serve as the first responders at the scene of incidents and emergencies
  Interventions: Other: Survey by Questionnaire

INTERVENTIONS:
Other: Survey by Questionnaire — The questionnaire is designed to collect the following information: demographic data (including gender, age, education level, marital status, place of residence, and whether the respondent is a healthcare provider), the respondent's status of basic life support (BLS) training, attitudes and willingness to use an automated external defibrillator (AED), and their knowledge of emergency medical service regulations.

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) remains a time-critical emergency where early cardiopulmonary resuscitation (CPR) and timely defibrillation using an automated external defibrillator (AED) are key to improving survival and neurological outcomes. Although Taipei has implemented dispatch-assisted CPR, delays remain between arrest recognition and AED application due to manpower and policy limitations. International guidelines, including the Global Resuscitation Alliance's ten steps to improve OHCA outcomes, recommend involving police as first responders. Prior studies from the United States and Switzerland demonstrate that police often arrive before emergency medical services (EMS), underscoring their potential role in reducing response times. However, police have not been officially included in OHCA dispatch systems in any region of Taiwan. This study aims to evaluate the willingness of police officers in New Taipei City to participate in prehospital resuscitation through a structured questionnaire. The survey also explores perceived facilitators and barriers to involvement. Findings will inform future training programs and strategies to promote police integration into prehospital emergency response systems, with the ultimate goal of improving OHCA survival rates.

DETAILED DESCRIPTION:
For patients with emergency cardiopulmonary arrest before arriving at the hospital, every second counts, especially good early cardiopulmonary resuscitation (Cardiopulmonary Resuscitation, CPR) and early use of automated external defibrillator (Automated External Defibrillator, referred to as AED), which can increase the patient's recovery of autonomous cardiopulmonary opportunity to cycle. After the introduction of online Dispatch-assisted CPR from Taipei, the survival rate and the rate of discharge with good neurology improved. Unfortunately, due to the limitations of manpower space and policies, the proportion and time from the successful identification of cardiopulmonary arrest to the first use of public electric shock is still relatively long. Ten guidelines recommended by the Global Resuscitation Alliance to improve survival for patients with pre-hospital cardiac arrest also recommend including police as first responders. Through more intensive manpower distribution, response times and shock times can be reduced, and these advances have also successfully improved survival rates. According to studies in the United States and Switzerland in 2002 and 2017, respectively, the police arrived at the scene faster than the emergency medical technician, which is also in line with the purpose of reducing reaction time and improving the survival rate of patients. No county or city in Taiwan has officially included the police in the OHCA dispatch. This study uses a questionnaire survey to understand the New Taipei City police's willingness to participate in the first aid and resuscitation of patients with cardiopulmonary arrest before hospitalization. At the same time, we will further analyze and understand the assistance and resistance of participating in emergency resuscitation. After the study is completed, courses such as education and training will be designed according to the results, and efforts will be made to reduce resistance, so that the police can be more involved in pre-hospital emergency resuscitation, in order to further improve the survival chances of patients with pre-hospital cardiopulmonary arrest.

ELIGIBILITY:
Inclusion Criteria:

* New Taipei City Government Police

Exclusion Criteria:

* Those who are unwilling to fill out this questionnaire or feel physically or mentally unwell while filling it out

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Frontline Police Officers in New Taipei City
Sampling Method: Non-Probability Sample
Enrollment: 4867 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Willingness to Perform CPR and Use an AED at the Scene of an Emergency | Baseline
  This outcome assesses whether participants are willing to go to the scene of an emergency under the command of the duty center to directly perform CPR and use AED to help patients. Options include: Yes; No.
Willingness to Receive AED Location Notification and Assist in Delivery and Use | Baseline
  This outcome assesses whether participants are willing to receive alerts from the dispatch center about nearby AED locations and assist in delivering the AED to the emergency scene and using it. Options include: Yes; No.

SECONDARY OUTCOMES:
Sex | Baseline
  This outcome evaluates responses to the question: "Gender." Options include: Male; Female.
Year of Birth | Baseline
  This outcome collects data on the participant's year of birth. This is a numerical, free-text entry used to assess age distribution.
Education Level | Baseline
  This outcome evaluates participants' highest attained level of education. Options include: High school; College or vocational school; Master's degree; Doctoral degree.
Marital Status | Baseline
  This outcome assesses the participant's marital status. Options include: Single; Married; Divorced.
Years of Service | Baseline
  This outcome collects data on the participant's length of service. Participants are asked to specify their years of service in both administrative and frontline (field) positions.
Co-residence with Elderly | Baseline
  This outcome evaluates whether participants live with adults aged 65 or older. Options include: Yes - number of people; No.
Awareness of AED | Baseline
  This outcome assesses whether participants have heard of an Automated External Defibrillator (AED). Options include: Yes; No.
Ability to Identify AED in Public | Baseline
  This outcome investigates whether participants believe they can identify an AED in a public setting. Options include: Yes; No.
Willingness to Use CPR + AED in Emergencies | Baseline
  This outcome evaluates the participant's willingness to perform cardiopulmonary resuscitation (CPR) and use an AED during emergencies. Options include: Yes; No.
Concerns About Performing CPR + AED (Multiple Selection) | Baseline
  This outcome identifies concerns participants may have about performing CPR and using an AED. Options include:
  1. Concern about legal or medical liability
  2. Concern about lack of skills causing harm
  3. Never seen an AED
  4. Belief that only trained personnel should use AEDs
  5. Other (please specify)
Confidence in Performing CPR | Baseline
  This outcome evaluates whether participants feel confident in their ability to perform CPR. Options include: Yes; No.
Confidence in Using AED | Baseline
  This outcome evaluates whether participants feel confident in their ability to use an AED. Options include: Yes; No.
Belief in Ability to Accurately Perform CPR | Baseline
  This outcome assesses whether participants believe they can accurately perform CPR. Options include: Yes; No.
Belief in Ability to Accurately Use AED | Baseline
  This outcome assesses whether participants believe they can accurately use an AED. Options include: Yes; No.
Previous Training in CPR + AED | Baseline
  This outcome assesses whether the participant has ever received training related to CPR and AED use. Options include: Yes; No.
Timing of Most Recent CPR + AED Training | Baseline
  This outcome evaluates the recency of the participant's latest CPR and AED training. Options include:
  1. Within the past 6 months
  2. Between 6 months and 1 year
  3. More than 1 year ago
  4. Never received training
Type and Duration of Last Training | Baseline
  This outcome assesses the format and total duration (in hours) of the participant's most recent CPR + AED training. Options include:
  1. In-person training
  2. Online training
  3. Blended (online + in-person) Total training hours: (open entry)
Perceived Eligibility to Use AED | Baseline
  This outcome evaluates who participants believe is eligible to use an AED. Options include:
  1. Medical personnel
  2. Emergency medical responders
  3. Staff at AED-installed locations
  4. Anyone capable of using it
  5. Not sure
Willingness to Use CPR + AED on Strangers | Baseline
  This outcome evaluates participants' willingness to perform CPR and use an AED on strangers. Options include: Yes; No.
Reasons for Unwillingness to Perform CPR + AED on Strangers (Multiple Selection) | Baseline
  This outcome identifies reasons why participants may be unwilling to assist strangers. Options include:
  1. Concern about legal or medical liability
  2. Concern about lack of skills causing harm
  3. Belief AEDs should be used only by trained personnel
  4. Unfamiliar with CPR or AED
  5. Prefer to assist only family or friends
  6. Concern about hygiene or infectious diseases
  7. Other (please specify)
Belief that the Public Should Learn CPR + AED | Baseline
  This outcome assesses whether participants believe all citizens should be trained in CPR and AED use. Options include: Yes; No; Other (please specify).
Willingness to Attend Free CPR + AED Course | Baseline
  This outcome evaluates whether participants are willing to attend a free CPR and AED training course. Options include: Yes; No.
Willingness to Spend Time on Free CPR + AED Course | Baseline
  This outcome assesses how much time participants are willing to spend attending a free CPR + AED course. Options include:
  1. Less than 1 hour
  2. 1 to 2 hours
  3. 2 to 3 hours
  4. 3 to 4 hours
  5. More than 4 hours
Main Reason for Not Attending Free CPR + AED Course | Baseline
  This outcome identifies the main reason participants are not willing to attend a free CPR and AED course. Options include:
  1. I don't need it
  2. I have a full schedule
  3. I already receive regular CPR + AED training
  4. Other (please specify)
Awareness of Good Samaritan Law | Baseline
  This outcome evaluates whether participants have heard of the Good Samaritan Law. Options include: Yes; No.
Impact of Good Samaritan Law on Willingness to Perform CPR + AED | Baseline
  This outcome evaluates whether knowledge of the Good Samaritan Law increases participants' willingness to perform CPR and use an AED. Options include: Yes; No.
Reasons for Unwillingness to Deliver and Use an AED (Multiple Selection) | Baseline
  This outcome identifies the reasons why participants may be unwilling to deliver and use an AED during an emergency. Options include:
  1. Concern about legal or medical liability
  2. Concern about lack of skills causing further harm
  3. Belief that AEDs should only be used by trained emergency responders
  4. I have never seen an AED
  5. I would prefer to use it only on family or friends
  6. I believe it is the fire department's responsibility
  7. I do not want to increase my workload
Incentives That May Increase Willingness to Deliver and Use an AED (Multiple Selection) | Baseline
  This outcome evaluates potential incentives that could increase participants' willingness to deliver an AED to the scene and use it. Options include:
  1. Comprehensive education and training
  2. Legal or medical liability exemption
  3. Administrative rewards (e.g., commendation or merit award) if the patient recovers and is discharged
  4. Monetary rewards if the patient recovers and is discharged
  5. Other (please specify)
Reasons for Unwillingness to Perform CPR and Use an AED at the Scene (Multiple Selection) | Baseline
  This outcome identifies the reasons why participants may be unwilling to perform CPR or use an AED at the scene of an emergency. Options include:
  1. Concern about legal or medical liability
  2. Concern about insufficient skills causing harm
  3. Belief that CPR should only be performed by trained emergency personnel
  4. I do not know how to perform CPR
  5. I would prefer to assist only family or friends
  6. I believe this is the fire department's responsibility
  7. I do not want to increase my workload
Incentives That May Increase Willingness to Perform CPR and Use an AED at the Scene (Multiple Selection) | Baseline
  This outcome evaluates potential factors that may increase participants' willingness to perform CPR and use an AED at the scene of an emergency. Options include:
  1. Comprehensive education and training
  2. Legal or medical liability exemption
  3. Administrative rewards (e.g., commendation or merit award) if the patient recovers and is discharged
  4. Monetary rewards if the patient recovers and is discharged
  5. Other (please specify)
Perceived Effectiveness of Police Administering CPR and AED Before EMS Arrival | Baseline
  This outcome assesses whether participants believe that police officers performing CPR and using an AED before the fire department or EMS arrives can help the patient. Options include:
  1. Yes, I believe it can help
  2. No, I do not believe it can help

CONTACTS AND LOCATIONS:
Overall Officials: Jen Tang Sun, Chief of Emergency Surgery, Study Chair — Far Eastern Memorinal Hospital
Locations (1):
- Far Eastern Memorinal Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Personal privacy protection

REFERENCES:
- [Background] Stein P, Spahn GH, Muller S, Zollinger A, Baulig W, Bruesch M, Seifert B, Spahn DR. Impact of city police layperson education and equipment with automatic external defibrillators on patient outcome after out of hospital cardiac arrest. Resuscitation. 2017 Sep;118:27-34. doi: 10.1016/j.resuscitation.2017.06.017. Epub 2017 Jun 24. PMID 28655625
- [Background] Krammel M, Lobmeyr E, Sulzgruber P, Winnisch M, Weidenauer D, Poppe M, Datler P, Zeiner S, Keferboeck M, Eichelter J, Hamp T, Uray T, Schnaubelt S, Nuernberger A. The impact of a high-quality basic life support police-based first responder system on outcome after out-of-hospital cardiac arrest. PLoS One. 2020 Jun 2;15(6):e0233966. doi: 10.1371/journal.pone.0233966. eCollection 2020. PMID 32484818
- [Background] Myerburg RJ, Fenster J, Velez M, Rosenberg D, Lai S, Kurlansky P, Newton S, Knox M, Castellanos A. Impact of community-wide police car deployment of automated external defibrillators on survival from out-of-hospital cardiac arrest. Circulation. 2002 Aug 27;106(9):1058-64. doi: 10.1161/01.cir.0000028147.92190.a7. PMID 12196329
- [Background] Hawkes C, Booth S, Ji C, Brace-McDonnell SJ, Whittington A, Mapstone J, Cooke MW, Deakin CD, Gale CP, Fothergill R, Nolan JP, Rees N, Soar J, Siriwardena AN, Brown TP, Perkins GD; OHCAO collaborators. Epidemiology and outcomes from out-of-hospital cardiac arrests in England. Resuscitation. 2017 Jan;110:133-140. doi: 10.1016/j.resuscitation.2016.10.030. Epub 2016 Nov 17. PMID 27865775
- [Background] Colquhoun MC, Chamberlain DA, Newcombe RG, Harris R, Harris S, Peel K, Davies CS, Boyle R. A national scheme for public access defibrillation in England and Wales: early results. Resuscitation. 2008 Sep;78(3):275-80. doi: 10.1016/j.resuscitation.2008.03.226. Epub 2008 Jun 17. PMID 18562074
- [Background] Rea TD, Olsufka M, Bemis B, White L, Yin L, Becker L, Copass M, Eisenberg M, Cobb L. A population-based investigation of public access defibrillation: role of emergency medical services care. Resuscitation. 2010 Feb;81(2):163-7. doi: 10.1016/j.resuscitation.2009.10.025. Epub 2009 Dec 3. PMID 19962225
- [Background] Moore MJ, Hamilton AJ, Cairns KJ, Marshall A, Glover BM, McCann CJ, Jordan J, Kee F, Adgey AA. The Northern Ireland Public Access Defibrillation (NIPAD) study: effectiveness in urban and rural populations. Heart. 2008 Dec;94(12):1614-9. doi: 10.1136/hrt.2007.130534. Epub 2008 Jan 29. PMID 18230637
- [Background] Blom MT, Beesems SG, Homma PC, Zijlstra JA, Hulleman M, van Hoeijen DA, Bardai A, Tijssen JG, Tan HL, Koster RW. Improved survival after out-of-hospital cardiac arrest and use of automated external defibrillators. Circulation. 2014 Nov 18;130(21):1868-75. doi: 10.1161/CIRCULATIONAHA.114.010905. PMID 25399395
- [Background] Pei-Chuan Huang E, Chiang WC, Lu TC, Wang CH, Sun JT, Hsieh MJ, Wang HC, Yang CW, Lin CH, Lin JJ, Yang MC, Huei-Ming Ma M. Barriers to bystanders defibrillation: A national survey on public awareness and willingness of bystanders defibrillation☆. J Formos Med Assoc. 2021 Mar;120(3):974-982. doi: 10.1016/j.jfma.2020.10.020. Epub 2020 Nov 18. PMID 33218851
- [Background] Kitamura T, Iwami T, Kawamura T, Nagao K, Tanaka H, Hiraide A; Implementation Working Group for the All-Japan Utstein Registry of the Fire and Disaster Management Agency. Nationwide public-access defibrillation in Japan. N Engl J Med. 2010 Mar 18;362(11):994-1004. doi: 10.1056/NEJMoa0906644. PMID 20237345